CLINICAL TRIAL: NCT04978584
Title: Smart Stop: A Phase II Trial of Rituximab, Lenalidomide, Acalabrutinib, Tafasitamab Prior to and With Standard Chemotherapy for Patients With Newly Diagnosed DLBCL
Brief Title: Rituximab, Lenalidomide, Acalabrutinib, Tafasitamab Alone and With Combination Chemotherapy for the Treatment of Newly Diagnosed Non-germinal Center Diffuse Large B-Cell Lymphoma, Smart Stop Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0046; NCI-2021-04298 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0046 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-10; First posted 2021-07-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — acalabrutinib; Cyclophosphamide; Doxorubicin; Lenalidomide; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; tafasitamab; Immunoglobulins; Disulfides; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (uLTRA, CHOP) (Experimental): COHORT I (SMART STOP): Patients receive rituximab IV over 4-6 hours on day 1, acalabrutinib PO BID on days 1-21, lenalidomide QD on days 1-10, and tafasitamab IV over 2 hours on days 1, 8, and 15. Treatments repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  COHORT II (uLTRA-CHOP): Patients who achieve a complete response to the Smart Stop in Cohort I, receive rituximab IV over 4-6 hours on day 1, acalabrutinib PO BID on days 1-21, lenalidomide QD on days 1-10, and tafasitamab IV over 2 hours on days 1, 8, and 15. Treatments repeat every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive cyclophosphamide IV over 1 hour, doxorubicin hydrochloride IV over 15 minutes, vincristine IV over 15 minutes on day 1, and prednisone PO QD on days 1-5. Treatments repeat every 21 days for up to 6 cycles in the absence of disease progr
  Interventions: Drug: Acalabrutinib; Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Lenalidomide; Drug: Prednisone; Biological: Rituximab; Biological: Tafasitamab; Drug: Vincristine

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Biological: Tafasitamab — Given IV
  Other Names: Immunoglobulin, Anti-(Human Cd19 Antigen) (Human-mus musculus Monoclonal MOR00208 Heavy Chain), Disulfide with Human-mus musculus Monoclonal MOR00208 .Kappa.-chain, Dimer; Monjuvi; MOR-00208; MOR00208; MOR208; Tafasitamab-cxix; XmAb5574
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine

SUMMARY:
This phase II trial studies the effect of rituximab, lenalidomide, acalabrutinib, tafasitamab alone and in combination with chemotherapy in treating patients with newly diagnosed non-germinal center diffuse large B-cell lymphoma. Rituximab and tafasitamab are monoclonal antibodies that may interfere with the ability of tumor cells to grow and spread. Acalabrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as lenalidomide, cyclophosphamide, doxorubicin, and vincristine, and work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Anti-inflammatory drugs, such as prednisone lower the body's immune response and are used with other drugs in the treatment of some types of cancer. Giving rituximab, lenalidomide, acalabrutinib, tafasitamab alone and with combination chemotherapy may help control non-germinal center diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate at the end of 4 cycles of therapy with rituximab, lenalidomide, acalabrutinib, tafasitamab in patients with high risk newly diagnosed non-germinal center B-cell (GCB) diffuse large B-cell lymphoma (DLBCL).

II. To determine the complete response rate at the end of 10 cycles of therapy with rituximab, lenalidomide, acalabrutinib, tafasitamab and chemotherapy (cyclophosphamide-hydroxydaunorubicin-oncovin-prednisone [CHOP]) in patients with high risk newly diagnosed non-GCB DLBCL.

SECONDARY OBJECTIVES:

I. To determine the overall response rate, survival outcomes (progression free and overall survival), and safety of rituximab, lenalidomide, acalabrutinib, tafasitamab and chemotherapy (CHOP) in patients with high risk newly diagnosed non-GCB DLBCL.

II. To evaluate the outcomes of patients who receive 10 cycles of rituximab, lenalidomide, acalabrutinib, tafasitamab with 6 concurrent cycles of CHOP in contrast to patients who receive a response adapted 2 concurrent cycles of CHOP in cohort 1.

III. To evaluate the outcomes of patients who receive 10 cycles of rituximab, lenalidomide, acalabrutinib, tafasitamab with 6 concurrent cycles of CHOP in contrast to patients who receive a response adapted 0 concurrent cycles of CHOP in cohort 2.

EXPLORATORY OBJECTIVE:

I. To evaluate the baseline and therapy induced changes in the profile of mutations, gene expression, minimal residual disease circulating tumor deoxyribonucleic acid (ctDNA) levels, immune cell subsets, in patients with newly diagnosed non-GCB DLBCL.

OUTLINE:

COHORT I (SMART STOP): Patients receive rituximab intravenously (IV) over 4-6 hours on day 1, acalabrutinib orally (PO) twice daily (BID) on days 1-21, lenalidomide once daily (QD) on days 1-10, and tafasitamab IV over 2 hours on days 1, 8, and 15. Treatments repeat every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

COHORT II (uLTRA-CHOP): Patients who achieve a complete response to the Smart Stop in Cohort I, receive rituximab IV over 4-6 hours on day 1, acalabrutinib PO BID on days 1-21, lenalidomide QD on days 1-10, and tafasitamab IV over 2 hours on days 1, 8, and 15. Treatments repeat every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive cyclophosphamide IV over 1 hour, doxorubicin hydrochloride IV over 15 minutes, vincristine IV over 15 minutes on day 1, and prednisone PO QD on days 1-5. Treatments repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve less than a complete response, receive rituximab IV over 4-6 hours on day 1, acalabrutinib PO BID on days 1-21, lenalidomide QD on days 1-10, and tafasitamab IV over 2 hours on days 1, 8, and 15. Patients also receive cyclophosphamide IV over 1 hour, doxorubicin hydrochloride IV over 15 minutes, vincristine IV over 15 minutes on day 1, and prednisone PO QD on days 1-5. Treatments repeat every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, then every 4 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed diagnosis of DLBCL.
2. No prior treatment except a prior limited-field radiotherapy, a short course of glucocorticoids ≤50mg daily of prednisone equivalent which must be no more than 4 days in duration and cease prior to day 1 of cycle 1, and/or 1 dose of cyclophosphamide 750mg/m2 for an urgent lymphoma related problem at diagnosis (e.g. epidural cord compression, superior vena cava syndrome).
3. Age ≥ 18 years and able to provide informed consent.
4. Participants must have bi-dimensional measurable disease, as defined as radiographically apparent disease with the longest dimension of ≥1.5cm.
5. Participants with performance status of ≤3 (3 only allowed if decline in status is deemed related to lymphoma and felt potentially reversible by the treating physician).
6. Serum bilirubin <1.5x ULN except in participants with Gilbert's syndrome as defined by > 80% unconjugated bilirubin who must have a serum bilirubin of <4x ULN; AST (SGOT) and ALT (SGPT) ≤ 3x ULN or < 5x ULN if hepatic metastases are present; ANC >1000/mm3 and platelets >100,000/mm3 unless deemed related to lymphoma involvement in the bone marrow and felt potentially reversible by the treating physician.
7. Renal function assessed by calculated creatinine clearance:

   a. Calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula. See section below, "Dosing Regimen", regarding lenalidomide dose adjustment for calculated creatinine clearance ≥ 30ml/min and < 60ml/min.
8. Participants must be willing to receive transfusions of blood products.
9. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
10. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
11. Women of childbearing potential and men who are sexually active with a woman of childbearing potential must be practicing a highly effective method of during and after the study (12 months after study drug for women and 3 months after study drug for men), consistent with local regulations regarding the use of birth control methods for participants participating in this clinical study. Men must agree to not donate sperm during and for up to 3 months after their conclusion of therapy on study.
12. Able to take aspirin (81 mg) daily or alternative therapy as prophylactic anticoagulation

Exclusion Criteria:

1. Any serious medical condition including but not limited to uncontrolled hypertension, uncontrolled congestive heart failure within past 6 months prior to screening (Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification), uncontrolled or symptomatic arrhythmias with corrected QT interval (QTc) > 480 msec at screening, uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, COPD, LVEF less than 40%, renal failure, uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura active infection, history of invasive fungal infection, moderate to severe hepatic disease (Child Pugh Class B or C), active hemorrhage, laboratory abnormality, or psychiatric illness that, in the investigators opinion places the participant at unacceptable risk and would prevent the subject from signing the informed consent form. Participants with history of cardiac arrhythmias should have cardiac evaluation and clearance.
2. Pregnant or lactating females.
3. Known hypersensitivity to lenalidomide or thalidomide, acalabrutinib, tafasitamab, rituximab, vincristine, doxorubicin, cyclophosphamide, or prednisone.
4. Known HIV infection. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative DNA polymerase chain reaction (PCR) and must be willing to undergo DNA PCR testing during the study to be eligible. Those who are HBsAg positive or hepatitis B DNA PCR positive will be excluded. Participants who are hepatitis C antibody positive will need to have a negative DNA PCR result to be eligible. Those who are hepatitis C DNA PCR positive will be excluded.
5. All participants with known central nervous system involvement with lymphoma.
6. Diagnosis of prior malignancy within the past 2 years with the exception of successfully treated basal cell carcinoma, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast. History of other malignancies are allowed if in remission (including prostate cancer participants in remission from radiation therapy, surgery or brachytherapy), not actively being treated, with a life expectancy > 3 years.
7. Significant neuropathy (Grades 2 or Grade 1 with pain) within 14 days prior to enrollment
8. Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis not due to lymphoma.
9. Participants with active pulmonary embolism or deep vein thrombosis (diagnosed within 30 days of study enrollment).
10. Participants with severe bradycardia (heart rate <40 bpm, hypotension, light-headedness, syncope).
11. Major surgery within 4 weeks of study entry, or wound that is not healed from prior surgery or trauma.
12. History of stroke or intracranial hemorrhage within 6 months prior to study entry.
13. Requires anticoagulation with warfarin or equivalent vitamin K antagonists.
14. Requires chronic treatment with strong CYP3A inhibitors.
15. Vaccinated with live, attenuated vaccines within 4 weeks of study entry.
16. Active bleeding or history of bleeding diathesis (eg, hemophilia or von Willebrand disease).
17. Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
18. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
19. Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) >2x ULN.
20. Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Note: Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
21. Concurrent participation in another therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2027-01-16 (Estimated); Study Completion 2027-01-16 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | At the end of 4 cycles of therapy with rituximab, lenalidomide, acalabrutinib, tafasitamab (each cycle = 21 days)
  The response rate and exact 95% confidence intervals will be calculated.
Complete response rate | At the end of 10 cycles of therapy with rituximab, lenalidomide, acalabrutinib, tafasitamab and chemotherapy (each cycle = 21 days)
  The response rate and exact 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 30 days post-treatment
  The unacceptable toxicity rate and exact 95% confidence intervals will be calculated. AE data will be summarized by frequency tables for all patient
Progression free survival | From study entry to objective disease progression or death from any cause, whichever occurs first, assessed up to 2 years post-treatment
  Will be estimated using the method of Kaplan and Meier.
Overall survival | Time between study entry and death from any cause, assessed up to 2 years post-treatment
  Will be estimated using the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Westin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Westin J, Davis RE, Feng L, Hagemeister F, Steiner R, Lee HJ, Fayad L, Nastoupil L, Ahmed S, Rodriguez A, Fanale M, Samaniego F, Iyer SP, Nair R, Oki Y, Fowler N, Wang M, Ma MCJ, Vega F, McDonnell T, Pinnix C, Griffith D, Lu Y, Tewari S, Sun R, Scott DW, Flowers CR, Neelapu S, Green MR. Smart Start: Rituximab, Lenalidomide, and Ibrutinib in Patients With Newly Diagnosed Large B-Cell Lymphoma. J Clin Oncol. 2023 Feb 1;41(4):745-755. doi: 10.1200/JCO.22.00597. Epub 2022 Aug 11. PMID 35952327
- See also: MD Anderson Cancer Center — http://www.mdanderson.org